CLINICAL TRIAL: NCT03023436
Title: Cytoreductive Surgery Combined With Hyperthermic Intraperitoneal Chemotherapy and Systemic Chemotherapy in Gastric Cancer With Regional Peritoneal Metastasis, a Multicenter and Single-arm Phase III Study
Brief Title: Cytoreductive Surgery Combined With HIPEC and Chemotherapy for Gastric Cancer With Peritoneal Metastasis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Guoxin Li, Principal Investigator, Nanfang Hospital, Southern Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLASS - 05
Record Dates: First submitted 2017-01-09; First posted 2017-01-18 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Stomach Neoplasm
Keywords: Stomach Neoplasms; Cytoreduction Surgical Procedures
MeSH Terms: conditions — Stomach Neoplasms | interventions — Cytoreduction Surgical Procedures; Hyperthermic Intraperitoneal Chemotherapy; Fluorouracil; Capecitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CRS + HIPEC + Systemic Chemotherapy (Experimental): Cytoreductive surgery(CRS) followed by Hyperthermic Intraperitoneal Chemotherapy(HIPEC) and systemic chemotherapy will be performed for the treatment of patients assigned to this group.
  CF regimens or other first line regimens based on Fluoropyrimidine and Cisplatin according to the National Comprehensive Cancer Network（NCCN） Guidelines （Gastric Cancer，version 3.2016) are recommended.Regimens and dosing schedules are not limited in this trial.
  Interventions: Procedure: Cytoreductive surgery; Procedure: Hyperthermic Intraperitoneal Chemotherapy; Drug: Fluoropyrimidine; Drug: Cisplatin

INTERVENTIONS:
Procedure: Cytoreductive surgery — Gastrectomy with D2 lymph node dissection and Metastasectomy for peritoneal metastatic sites only.
  A total, distal, or proximal gastrectomy and the type of reconstruction will be selected according to the surgeon's experience.
  Metastasectomy is limited to peritoneal metastatic sites only to render the patient no evidence of disease (NED) with at least 1cm negative margins when possible.
  Other Names: CRS , Cytoreduction Surgical Procedures
Procedure: Hyperthermic Intraperitoneal Chemotherapy — Docetaxel 120 mg diluted in 5.0 L of saline is forced into the abdomen through the inflow catheter by a pump and pulled out through the drains as a heated intraperitoneal perfusion.A heat exchanger keeps the intraperitoneal fluid at 43±0.5℃ and duration limited to 70 minutes.24 hours after cytoreductive surgery no less than 2 cycles postoperative chemotherapy will be recommended.
  Other Names: HIPEC
Drug: Fluoropyrimidine — CF regimens or other first line regimens based on Fluoropyrimidine and Platinum according to the NCCN Guidelines（Gastric Cancer，version 3.2016) are recommended.Regimens and dosing schedules are not limited in this trial.
  Other Names: fluorouracil or capecitabine
Drug: Cisplatin — CF regimens or other first line regimens based on Fluoropyrimidine and Platinum according to the NCCN Guidelines（Gastric Cancer，version 3.2016) are recommended.Regimens and dosing schedules are not limited in this trial.
  Other Names: cis-diamine dichloroplatinum(CDDP)

SUMMARY:
This study evaluates the survival benefit and safety of cytoreductive surgery(CRS) combined with HIPEC and chemotherapy in gastric cancer with peritoneal metastasis.

DETAILED DESCRIPTION:
Peritoneal metastasis is one of the most frequent non-curable factors in advanced gastric cancer with poor prognosis, the median survival time of patients is less than 1 year and even worse in China. Recently, several new modalities have been developed and reported to improve survival, including the new chemotherapeutic agents, molecular targeting agents and hyperthermic intraperitoneal chemotherapy（HIPEC）.Still, the long-term outcomes based on multicenter randomized clinical trials (RCTs) are awaited.

The surgical approach to metastatic lesions has been proved to play a very crucial role in prolonging the survival of metastatic colorectal patients, which might be able to cure patients with the operation aiming at R0 resection. For patients with metastatic gastric cancer, surgical intervention of primary tumor and measurable metastatic lesion is technically feasible, while the survival benefit is controversial. Even though the REGATTA trial demonstrated that the removal of the primary tumor is not necessarily beneficial, the role of operation aiming at R0 resection combined with new regimens like HIPEC and new chemotherapeutic agents is still confusing and new categories of classification for metastatic gastric cancer based on the treatment response is needed.

In order to evaluate the survival benefit and safety of cytoreductive surgery(CRS) and HIPEC before beginning chemotherapy in gastric cancer with peritoneal metastasis, patients who fulfill the inclusion and exclusion criteria will be recruited in this study and receive CRS, HIPEC and chemotherapy. Chemotherapy regimen based on cisplatin and fluorouracil(CF) are recommended. Patients are followed up for 2 years and the safety and survival outcome will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age from over 18 to under 75 years
* Histologically proven primary gastric adenocarcinoma confirmed pathologically by endoscopic biopsy
* Diagnosed with clinical T1-4N0-3M1（distant metastases confined to peritoneum, P1）according to the American Joint Committee on Cancer(AJCC) Cancer Staging Manual Seventh Edition by laparoscopic exploration
* Localized peritoneal metastasis with peritoneal cancer index(PCI) less than 20
* Resection of primary tumor and metastasis is anticipated to reach the CC0 status(no residual tumor )
* Performance status of 0 or 1 on Eastern Cooperative Oncology Group(ECOG) scale
* Written informed consent

Exclusion Criteria:

* Adenocarcinoma of esophageal-gastric junction(AEG) that requires thoracotomy
* Distant metastases not confined to peritoneum, including liver (H1), para-aortic lymphnode (stations 16a1 and/or b2), lung, brain, bone and other organs
* Histologically proven Human epidermal growth factor receptor 2(HER2)-neu overexpressing adenocarcinoma
* History of previous neoadjuvant chemotherapy , radiotherapy or clinical trial treatment within 3 months
* Contraindication for anesthesia, surgery, chemotherapeutic agents or HIPEC
* Women of child-bearing potential who are pregnant or breastfeeding
* History of prior/other malignancies within the 5 years prior to enrollment
* Cerebrovascular accident occurred within 6 months (myocardial infarction, unstable angina, cerebral infarction, or cerebral hemorrhage)
* History of continuous systematic administration of corticosteroids within one month
* Requirement of simultaneous surgery for other disease
* Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer
* FEV1<50% of predicted values

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2016-01; Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
2-year Median survival time | 24 months
  The time point when the cumulative survival rate is 50% according to the survival curve.

SECONDARY OUTCOMES:
2-year overall survival rate | 24 months
  Overall survival rate calculated according to the survival curve.
Progression free survival rate | 24 months
  Progression free survival rate calculated according to the disease progression curve.
Morbidity and mortality | 30 days; 24 months
  The early complication and mortality are defined as the event observed within 30 days after intervention, while the time frame for late complication is the period beyond 30 days after intervention to the end of month 24th. Complications are ranked from grade 0-5 according to CTCAE V4.0

OTHER OUTCOMES:
Quality of life(site-specific module for gastric cancer) | Every 6 months to 2 years
  Evaluated according to European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Stomach(EORTC QLQ-STO22)
Quality of life | Every 6 months to 2 years
  Evaluated according to European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Cancer (EORTC QLQ-C30)
circulating tumor cell（CTC） alteration | Every 6 months to 2 years
circulating tumor DNA（ctDNA）alteration | Every 3 months to 2 years
Molecular biomarker alteration | Every 6 months to 2 years
  Molecular biomarker includes 14 genes（TP53, BAI1, THSD1, ARID2, KIAA2022, ERBB4, ZNF721, NT5E, PDE10A, CA1, NUMB, NBN, ZFYVE16 and NCAM1） according to the whole-exome sequencing results.

CONTACTS AND LOCATIONS:
Overall Officials: Guoxin Li, Principal Investigator — Chinese Laparoscopic Gastrointestinal Surgery Study (CLASS) Group; Nanfang Hospital, Southern Medical University, China
Locations (13):
- China (13):
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Cancer Center of Guangzhou Medical University, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Meizhou People's Hospital, Meizhou, Guangdong
  - Zhongshan City People Hospital, Zhongshan, Guangdong
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Cutsem E, Moiseyenko VM, Tjulandin S, Majlis A, Constenla M, Boni C, Rodrigues A, Fodor M, Chao Y, Voznyi E, Risse ML, Ajani JA; V325 Study Group. Phase III study of docetaxel and cisplatin plus fluorouracil compared with cisplatin and fluorouracil as first-line therapy for advanced gastric cancer: a report of the V325 Study Group. J Clin Oncol. 2006 Nov 1;24(31):4991-7. doi: 10.1200/JCO.2006.06.8429. PMID 17075117
- [Background] Koizumi W, Narahara H, Hara T, Takagane A, Akiya T, Takagi M, Miyashita K, Nishizaki T, Kobayashi O, Takiyama W, Toh Y, Nagaie T, Takagi S, Yamamura Y, Yanaoka K, Orita H, Takeuchi M. S-1 plus cisplatin versus S-1 alone for first-line treatment of advanced gastric cancer (SPIRITS trial): a phase III trial. Lancet Oncol. 2008 Mar;9(3):215-21. doi: 10.1016/S1470-2045(08)70035-4. Epub 2008 Feb 20. PMID 18282805
- [Background] Bang YJ, Van Cutsem E, Feyereislova A, Chung HC, Shen L, Sawaki A, Lordick F, Ohtsu A, Omuro Y, Satoh T, Aprile G, Kulikov E, Hill J, Lehle M, Ruschoff J, Kang YK; ToGA Trial Investigators. Trastuzumab in combination with chemotherapy versus chemotherapy alone for treatment of HER2-positive advanced gastric or gastro-oesophageal junction cancer (ToGA): a phase 3, open-label, randomised controlled trial. Lancet. 2010 Aug 28;376(9742):687-97. doi: 10.1016/S0140-6736(10)61121-X. Epub 2010 Aug 19. PMID 20728210
- [Background] Fujitani K, Yang HK, Mizusawa J, Kim YW, Terashima M, Han SU, Iwasaki Y, Hyung WJ, Takagane A, Park DJ, Yoshikawa T, Hahn S, Nakamura K, Park CH, Kurokawa Y, Bang YJ, Park BJ, Sasako M, Tsujinaka T; REGATTA study investigators. Gastrectomy plus chemotherapy versus chemotherapy alone for advanced gastric cancer with a single non-curable factor (REGATTA): a phase 3, randomised controlled trial. Lancet Oncol. 2016 Mar;17(3):309-318. doi: 10.1016/S1470-2045(15)00553-7. Epub 2016 Jan 26. PMID 26822397
- [Result] Hu Y, Huang C, Sun Y, Su X, Cao H, Hu J, Xue Y, Suo J, Tao K, He X, Wei H, Ying M, Hu W, Du X, Chen P, Liu H, Zheng C, Liu F, Yu J, Li Z, Zhao G, Chen X, Wang K, Li P, Xing J, Li G. Morbidity and Mortality of Laparoscopic Versus Open D2 Distal Gastrectomy for Advanced Gastric Cancer: A Randomized Controlled Trial. J Clin Oncol. 2016 Apr 20;34(12):1350-7. doi: 10.1200/JCO.2015.63.7215. Epub 2016 Feb 22. PMID 26903580
- [Result] Geng X, Liu H, Lin T, Hu Y, Chen H, Zhao L, Mou T, Qi X, Yu J, Li G. Survival benefit of gastrectomy for gastric cancer with peritoneal carcinomatosis: a propensity score-matched analysis. Cancer Med. 2016 Oct;5(10):2781-2791. doi: 10.1002/cam4.877. Epub 2016 Sep 20. PMID 27650694